CLINICAL TRIAL: NCT03125707
Title: German MPN-Registry for BCR-ABL 1-Negative Myeloid Neoplasms (Study Group Ulm)
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Frank Stegelmann, Principal Investigator Dr. med., University of Ulm
Other Study IDs: MPN Registry - Ulm
Record Dates: First submitted 2017-01-11; First posted 2017-04-24 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: BCR-ABL1-Negative Myeloid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Registry study

SUMMARY:
To register a large number of patients with the diagnosis of a BCR-ABL 1- negative myeloid neoplasm (according to WHO 2008 / 2016 classification) in participating centers

To store samples from all patients (e.g. bone marrow aspirate, peripheral blood, plasma, and buccal swap, skin biopsy samples in exceptional cases)

To perform morphologic and genetic analyses

To assess clinical characteristics and outcome data using a defined catalogue containing clinically relevant variables

To assess biological disease features and correlate with clinical outcome data (prognostic and predictive markers)

To assess quality of life

DETAILED DESCRIPTION:
To register a large number of patients with the diagnosis of a BCR-ABL 1- negative myeloid neoplasm (according to WHO 2008 / 2016 classification) in participating centers

To store samples from all patients (e.g. bone marrow aspirate, peripheral blood, plasma, and buccal swap, skin biopsy samples in exceptional cases)

To perform morphologic and genetic analyses

To assess clinical characteristics and outcome data using a defined catalogue containing clinically relevant variables

To assess biological disease features and correlate with clinical outcome data (prognostic and predictive markers)

To assess quality of life

ELIGIBILITY:
Inclusion Criteria:

Both female and male patients meeting the mentioned inclusion criteria will be included in this registry, because the risk to get a myeloid neoplasm does not depend on a patient's gender. Patients must meet all of the following inclusion criteria to be eligible for enrollment into the registry:

* Patients with BCR-ABL 1-myeloid neoplasia according to WHO classification or IWG MRI criteria
* Age ≥ 18 years. There is no upper age limit.
* Signed written informed consent.

Exclusion Criteria:

* Severe neurological or psychiatric disorder interfering with ability to give an informed consent
* No consent for registration, storage and handling of the personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of a BCR-ABL 1-negative myeloid neoplasm in participating centers
Sampling Method: Non-Probability Sample
Enrollment: 2172 (Estimated)
Dates: Start 2013-05; Primary Completion 2045-09 (Estimated); Study Completion 2045-09 (Estimated)

PRIMARY OUTCOMES:
Treatment decision | 25 years
  Treatment decision (watch and wait, standard, investigational)
Response | 25 years
  Response of treatment
Overall survival | 25 years
  Survival over the whole study duration
Progression-free-survival | 25 years
  Survival without any progression
Duration of response | 25 years
  Duration of response over the whole study duration
Quality of life assessed by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF Protocol 5/25/11, EORTC QLQ-C30, FACT-Lym (Fassung 4)), supplemented by information on self-assessed concomitant diseases and demographics. | 25 years
  Quality of life assessed by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF Protocol 5/25/11, EORTC QLQ-C30, FACT-Lym (Fassung 4)), supplemented by information on self-assessed concomitant diseases and demographics.

CONTACTS AND LOCATIONS:
Locations (30):
- Germany (30):
  - Hämatologische Onkologie Praxis Augsburg, Augsburg
  - Klinikum Augsburg, Augsburg
  - Helios Klinikum, Bad Saarow, Bad Saarow
  - Klinikum Mittelbaden, Baden-Baden
  - MVZ Klinikum Coburg, Coburg
  - Donauwörth, Onko-Medeor, Donauwörth
  - Onkologie, BAG, Dresden, Dresden
  - Onkologie Erding, Erding
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Alb Fils Kliniken Göppingen, Göppingen
  - Universitätsklinikum Greifswald, Greifswald
  - Onkologische Praxis, Heidelberg, Heidelberg
  - Onkologische Schwerpunktpraxis, Heilbronn, Heilbronn
  - Marienhospital Bochum-Herne, Herne
  - Universitätsklinikum Jena, Jena
  - Klinikum Kempten-Oberallgäu gGmbH, Kempten
  - Landshut VK&K Studien GbR, Landshut
  - Leer, Studienzentrum Unter Ems, Leer
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsklinikum Mannheim, Mannheim
  - Mannheim, Onkologiepraxis, Mannheim
  - Memmingen, Onkologiepraxis, Memmingen
  - Mühlenkreiskliniken Minden, Minden
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Stuttgart, MVZ am RBK, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Rems-Murr-Kliniken Winnenden, Winnenden
  - Würzburg / Kitzingen, Gemeinschaftspraxis Dr. Schlag, Würzburg

IPD SHARING:
Plan to Share IPD: No